CLINICAL TRIAL: NCT07167381
Title: xDRIVE Functional Precision Medicine + Artificial Intelligence Individualized Treatments for Florida-based Cancer Patients With Relapsed/ Refractory Cancers
Brief Title: xDRIVE for Florida-based Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Ascent Biomedical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAB00000002; Grant # 25C13 (Other Grant/Funding Number: Florida Cancer Innovation Fund - Florida Department of Health)
Record Dates: First submitted 2025-08-24; First posted 2025-09-11 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Cancer; Neoplams; Refractory; Recurrence; Leukaemia; Lymphoma; Solid Tumor Malignancies; Solid Cancers
Keywords: Functional Precision Medicine; Artificial Intelligence
MeSH Terms: conditions — Neoplasms; Recurrence; Leukemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- xDRIVE Profiling (Experimental): Patients will receive tumor profiling via xDRIVE Functional Precision Medicine and Artificial Intelligence analysis
  Interventions: Diagnostic Test: xDRIVE Tumor Profiling

INTERVENTIONS:
Diagnostic Test: xDRIVE Tumor Profiling — Patients and physicians will receive tumor profiling data via xDRIVE Functional Precision Medicine and Artificial Intelligence analysis. As this is a feasibility study, results will be returned to the physician and the physician may use the data to inform the next line of treatment.

SUMMARY:
Through this study funded by the Florida Cancer Innovation Fund, First Ascent will demonstrate state-wide feasibility of providing xDRIVE Functional Precision Medicine + Artificial Intelligence platform by assessing patient clinical benefit and health economics impacts. As this is a feasibility study, results will be returned to the physician and the physician may use the data to inform the next line of treatment. The investigator will run a prospective single-arm feasibility study providing the xDRIVE FPM AI platform to n = 210+ cancer patients throughout the state of Florida, especially those from underserved populations (pediatric patients and patients in Black, Brown, Hispanic, and rural communities).

DETAILED DESCRIPTION:
Cancer remains a leading cause of death in Florida, presenting formidable challenges across different patient populations resulting in over with 138,000 deaths in the previous 5 years. For children, cancer is the leading cause of death by disease, with pediatric malignancies often being particularly aggressive. Notably, 5-year overall survival rates for children with certain aggressive subtypes often fall below 30%. Similarly, adult cancer patients, especially those in minority and rural communities, face significant health and economic disparities that impede their access to care and contribute to poorer outcomes. For both pediatric and adult patients, these challenges are often compounded by systemic barriers, including insurance denials for potentially effective off-label drug use and the prohibitive cost of travel required to access specialized care at major cancer centers. To address these critical gaps, First Ascent is opening a clinical program, funded by the Florida Cancer Innovation Fund, that will provide cutting-edge personalized cancer treatment to cancer patients throughout Florida. The program will provide the xDRIVE Functional Precision Medicine (FPM) and Artificial Intelligence platform to serve both pediatric and adult patients, with a particular focus on ensuring access for underserved communities.

Results from the clinical feasibility study on advanced pediatric solid and hematological cancers (NCT03860376) recently published in Nature Medicine demonstrated that 21 of 24 patients (87.5%) enrolled in the clinical trial had actionable treatment recommendations returned within median 10 days. Additionally, 83% (5/6) of FPM-guided patients had >30% longer progression-free survival (PFS) compared to their own previous regimens, with a median 8.5-fold increase in PFS. In contrast, only 13% (1/8) patients in the physician's choice arm had >30% longer PFS. These ongoing clinical programs serving patients at Nicklaus Children's Hospital and Cleveland Clinic Florida have demonstrated the feasibility and clinical benefit of xDRIVE FPM, which has been extended to patients around Florida and around the country. Updated outcomes from the ongoing FPM studies demonstrate that 92% of patients receive individualized treatment recommendations, and 95% of patients receive clinical benefit from FPM-guided treatment, even in heavily-pretreated recurrent/refractory patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent/refractory cancer patients up to age 18 (willing to sign assent if ages 7 - 17 years)
* -OR- Patients with recurrent/refractory cancer ≥18 years of age.
* Patients who have received at least one prior line of standard of care therapy.
* Patients able to provide treatment and outcome information from previous line(s) of therapy.
* Patients with sufficient health status to undergo cancer therapy, e.g., Eastern Cooperative Group (ECOG) performance status of 0, 1, or 2 for adult patients.
* Patients who are scheduled for or have recently undergone a tumor biopsy, excision, or resection.
* Patients willing to have a blood draw or buccal swab performed for matched normal material for comparison during tumor DNA profiling.

Exclusion Criteria:

* Patients who do not have malignant tissue available and accessible, patients where the amount of excised malignant tissue is insufficient material for ex vivo drug testing and/or genetic profiling, defined as <0.3g for resections or core/fine-needle biopsies not containing malignant tissue by pathology review, or insufficient malignant tissue in peripheral blood or bone marrow aspirate samples.
* Patients with insufficient health indicators to undergo therapeutic intervention.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Return of treatment recommendations from xDRIVE functional precision medicine platform within a clinically-actionable timeframe | Return of xDRIVE data will be completed in under 2 weeks
  Tumor tissues provided by patients will undergo drug sensitivity testing and molecular tumor profiling in order to identify individualized treatment options. Treatment recommendations from both tumor profiling methods will be returned to the patient and physician to support clinical decision-making. Return of data in a timeframe fast enough to support decision-making is critical for showing clinical feasibility of this approach around the state of Florida. Feasibility will be demonstrated if xDRIVE treatment recommendations are returned within 2 weeks for at least 151 of 210 patients (72%), which is sufficient to reject the null hypothesis (≤60% of patients receiving treatment recommendations) with >95% power (α = 0.025).

SECONDARY OUTCOMES:
PFS Ratio ≥1.3x | 1 year after patient enrollment
  Progression-free survival (PFS) ratio ≥1.3x (ratio of program PFS vs. previous PFS) in patients guided by xDRIVE individualized treatments or by treatment of physician's choice. PFS ratio ≥1.3x in 30%+ of at least 62 patients, below our published rate of 83%, will provide >85% power (α = 0.025) to reject the null hypothesis (<15% PFS ratio ≥1.3).
Objective Response Rate (ORR) | 1 year after enrollment
  Objective responses in 45%+ in at least 76 patients, below our published 83% ORR, will provide >85% power (α = 0.025) to reject the null hypothesis (<30% ORR).
Disease Control Rate (DCR) | 1 year after enrollment
  Disease control in 62%+ in at least 76 patients will provide >85% power (α = 0.025) to reject the null hypothesis (<45% ORR).

OTHER OUTCOMES:
Rates of actionable treatments | Immediately following return of xDRIVE drug sensitivity testing and molecular tumor profiling data. Actionability will be tracked independent of treatment recommendations being returned within the 2 week timeframe for the primary objective
  Rates of actionable treatments from genomic tumor profiling versus xDRIVE profiling
Progression-free survival (PFS) | 1 year following enrollment
  Individual cancer types with sufficient patient enrollment and outcomes will be compared against historical PFS data
Overall Survival (OS) | 1 year following enrollment
  Individual cancer types with sufficient patient enrollment and outcomes will be compared against historical PFS data

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - First Ascent Biomedical, Miami, Florida
  - Florida International University, Miami, Florida

IPD SHARING:
Plan to Share IPD: Yes
Patient cancer types and relevant clinical outcomes data will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: If published, will be shared via open access publication.
Access Criteria: Data will be anonymized and will be published in open access journal. Access will be enabled through the publication and associated data

REFERENCES:
- [Background] Acanda de la Rocha AM, Berlow NE, Azzam DJ. Functional precision medicine: the future of cancer care. Trends Mol Med. 2025 May;31(5):404-408. doi: 10.1016/j.molmed.2024.10.015. Epub 2024 Nov 19. PMID 39567286
- [Background] Acanda De La Rocha AM, Berlow NE, Fader M, Coats ER, Saghira C, Espinal PS, Galano J, Khatib Z, Abdella H, Maher OM, Vorontsova Y, Andrade-Feraud CM, Daccache A, Jacome A, Reis V, Holcomb B, Ghurani Y, Rimblas L, Guilarte TR, Hu N, Salyakina D, Azzam DJ. Feasibility of functional precision medicine for guiding treatment of relapsed or refractory pediatric cancers. Nat Med. 2024 Apr;30(4):990-1000. doi: 10.1038/s41591-024-02848-4. Epub 2024 Apr 11. PMID 38605166